CLINICAL TRIAL: NCT02933450
Title: Relypsa For ED Acute Hyperkalemia Control and Reduction (REDUCE)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Relypsa, Inc. (Industry)
Responsible Party: Principal Investigator, Zubaid Rafique, Principal Investigator, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-39340
Record Dates: First submitted 2016-08-25; First posted 2016-10-14 (Estimated); Results first posted 2019-05-09 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Kidney Failure, Chronic
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — patiromer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patiromer group (Active Comparator): Patiromer 25.2 g dose
  Interventions: Drug: Patiromer 25.2 g
- Standard of Care group (No Intervention): Standard of Care

INTERVENTIONS:
Drug: Patiromer 25.2 g — Single dose of Patiromer 25.2 g
  Arms: Patiromer group

SUMMARY:
The Investigator hypothesize that a single dose of patiromer will lower serum potassium levels in less than 6hrs. Since a dosage of 30g/day for a period of 4 weeks has been studied in at least two multicenter randomized controlled trials, the Investigator further hypothesize that a single dose of 25.2g of patiromer will be well tolerated in hyperkalemic patients in the Emergency Department setting. The FDA approved dosage of 25.2g is appropriate for this study because the research staff will enroll patients with moderate (K greater than 6 mEq/L) to severe hyperkalemia, and the higher dosage has typically been used in this population for more effective control.

DETAILED DESCRIPTION:
This is an open label pilot study. Thirty patients with ESRD who qualify for emergent dialysis on the basis of serum potassium greater than 6mEq/L will be randomly assigned, using a random number generator in blocks of sixes, to standard-of-care (standard care) or patiromer group. Patients in the patiromer group will be given a single dose of 25.2g of patiromer in addition to standard-of-care treatment after randomization. Standard-of-care is defined as intervention or care provided by clinical provider according to individual practice pattern or hospital protocol. Each group of 15 patients will be observed with telemetry monitoring for 10 hours or till hemodialysis units become available for treatment (whichever comes first). Blood draws and electrocardiograms (ECGs) will be performed at enrollment and at 1, 2, 4, 6, 8 and 10hrs thereafter. Serum will be analyzed for basic metabolic panel and magnesium. Medications, including potassium lowering agents, administered during this period will be documented.

1. Informed consent will be obtained. 2. Subject will be randomized. 3. A. Randomized to Standard of Care (SOC): data will be collected on SOC treatment. 3. B. Randomized to patiromer group: subjects will receive a single dose of 25.2g of patiromer. SOC data will be collected. 4. all subjects will have blood drawn and ECGs (1 12 lead ECG and 1 Lead I Rhythm strip) done at baseline, 1, 2, 4, 6, 8 and 10 hours. Blood will be analyzed for basic metabolic panel and magnesium. 5. CRF completion-SOC data will be recorded in addition to current medications. 6. After subjects have received hemodialysis or reach the 10 hour study period, whichever comes first, the subject will be completed on the study.

ELIGIBILITY:
Inclusion Criteria:

* ESRD patients with serum potassium greater than or equal to 6.0 mEq/L
* Emergent dialysis not expected to be available for 6 hours

Exclusion Criteria:

* new clinically significant arrhythmia on initial ECG
* patiromer is contraindicated
* have received SPS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2016-08; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zubaid Rafique, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Ben Taub Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be coded and shared with the sponsor

RESULTS

PARTICIPANT FLOW:
Groups:
- Patiromer: Single dose of Patiromer 25.2 g + Standard of Care
- Standard of Care: Standard of Care
Period: Overall Study
Arm/Group | Patiromer | Standard of Care
Started | 20 | 23
Completed | 15 | 15
Not Completed | 5 | 8

BASELINE CHARACTERISTICS:
Groups:
- Patiromer Group: Single dose of Patiromer 25.2 g + Standard of Care
- Total: Total of all reporting groups
Arm/Group | Patiromer Group | Standard of Care Group | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 41 [36 to 50] | 48 [39 to 52] | 43 [36 to 52]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 13
  Male | 10 | 7 | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Patiromer in Reducing Serum Potassium
Description: serial serum potassium levels will be graphed and compared between the 2 groups
Time Frame: 6 hours
Measure: Mean (95% Confidence Interval); unit: mEq/L
Groups:
- Patiromer: Subjects receiving a single dose of Patiromer 25.2 g + Standard of Care therapy
- Standard of Care: subjects receiving standard of care therapy
Arm/Group | Patiromer | Standard of Care
Number analyzed (Participants) | 15 | 15
mEq/L
  1 hr | 6.17 [5.94 to 6.46] | 6.6 [6.33 to 6.86]
  2 hr | 5.9 [5.67 to 6.2] | 6.47 [6.21 to 6.73]
  4 hr | 5.73 [5.5 to 6.02] | 6.04 [5.77 to 6.30]
  6 hr | 5.81 [5.51 to 6.16] | 6.27 [5.97 to 6.58]

2. Secondary Outcome: Tolerability of High Dose Patiromer in ESRD Patients on Hemodialysis in the Acute Setting.
Description: adverse events will be recorded and compared between the 2 groups
Time Frame: 6 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Patiromer | Standard of Care
Number analyzed (Participants) | 14 | 15
Participants
  Total | 4 | 5
  GI side effects | 1 | 2
  Hypoglycemia | 3 | 3
  Hypomagnesemia | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected up to 6hrs
Arm/Group | Patiromer | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 4/15 | 5/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patiromer (N=15) | Standard of Care (N=15)
GI Side Effects (Gastrointestinal disorders) | 1 (1) | 2 (2) — Nausea, vomiting, diarrhea, constipation, abdominal bloating or pain
Hypoglycemia (General disorders) | 3 (3) | 3 (3) — Blood sugar < 70 mg/dL

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-21): https://cdn.clinicaltrials.gov/large-docs/50/NCT02933450/Prot_SAP_000.pdf